CLINICAL TRIAL: NCT01922180
Title: Chronic Obstructive Pulmonary Disease: CT Features of Severe Exacerbation
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Maxime HACKX, MD, Erasme University Hospital
Other Study IDs: COPD-EXAC-CT
Record Dates: First submitted 2013-08-09; First posted 2013-08-14 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: COPD Exacerbation
Keywords: Chest Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD Exacerbation: COPD patients aged 18 years or more, were included at the time of an exacerbation episode leading to admission in our hospital, which corresponds to a severe episode. There were no exclusion criteria. Patients underwent chest CT scans and PFT. After a minimum of two weeks free of any acute symptom after discharge, CT scans and PFT were redone.
  Interventions: Radiation: Chest CT scans

INTERVENTIONS:
Radiation: Chest CT scans — CT examinations were performed with a commercially available 64-detector row scanner. Images were acquired in supine position after full inspiration and full expiration, using the following parameters: slice thickness, 0.6 mm; pitch, 1.4; rotation time, 330 msec; tube voltage, 120 kiloVolts; and tube current-time product, 100 milliAmperes, with automatic exposure control (CareDose 4D, Siemens Healthcare) switched on. From raw data, 1-mm-thick section images were reconstructed at 0.7-mm intervals by using a high spatial algorithm and a soft-tissue algorithm. The inspiratory CT scan at the time of exacerbation was performed with intravenous iodinated contrast material, whereas the control scan was unenhanced.

SUMMARY:
To describe Computed Tomography (CT) features associated with severe exacerbations of Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
The natural course of COPD is associated with episodes of exacerbation which are clinically defined as acute events characterized by a worsening of the patient's respiratory symptoms that is beyond normal day-to-day variations and which leads to a change in medication. Moreover, these episodes can be classified into mild, moderate, or severe exacerbations, following patient's need for medical environment. While the cause of about one-third of severe exacerbation episodes cannot be identified, two-thirds are associated with certain conditions such as respiratory tract infections (viral or bacterial), air pollution, as well as pulmonary embolism (PE), pulmonary edema, cardiac arrhythmia, pneumothorax, or pleural effusion. As COPD exacerbations are associated with increased morbidity and mortality, as well as with increased healthcare costs, their prevention and treatment are two major objectives in COPD management with subsequent requirement for appropriate assessment tools. As imaging tool, chest radiography is limited to the detection of pneumonia and pleural abnormalities, and only leads to change in managements in a marginal proportion of patients. However, while Computed Tomography (CT) scans allows detecting more chest abnormalities, the knowledge of CT features at the time of exacerbation is a pre-requisite for determining possible role of CT in routine work-up of exacerbation. Nevertheless these features remain widely unknown, previous studies having focused on the prevalence of PE. The aim of our study was therefore to describe these features by comparing CT scans performed at severe exacerbation with control scans.

ELIGIBILITY:
Inclusion Criteria:

* Severe exacerbation episode of COPD, requiring hospital admission

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients followed in our institution (i.e. Erasme University Hospital), who are admitted for a severe exacerbation episode.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2007-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Chest CT scan features at exacerbation | 4 hours
  Grading the severity of the following 15 features: bronchiectasis, mucous plugging, bronchial wall thickening, pulmonary consolidation, ground glass opacity, cysts or bullae, air trapping, centrilobular micronodules, platelike atelectasis, emphysema, pulmonary embolism, pleural effusion, mediastinal or hilar lymphadenopathy, reticular pattern or honeycombing, and pulmonary mass or nodule.
Chest CT scan features at control | Minimum two weeks after exacerbation
  Grading the severity of the following 15 features: bronchiectasis, mucous plugging, bronchial wall thickening, pulmonary consolidation, ground glass opacity, cysts or bullae, air trapping, centrilobular micronodules, platelike atelectasis, emphysema, pulmonary embolism, pleural effusion, mediastinal or hilar lymphadenopathy, reticular pattern or honeycombing, and pulmonary mass or nodule.

SECONDARY OUTCOMES:
PFT at control | Minimum two weeks after exacerbation
  Measurements of the forced vital capacity (FVC), the forced expiratory volume in one second (FEV1), the functional residual capacity (FRC), the total lung capacity (TLC) and the residual volume (RV).
PFT at exacerbation | 4 hours
  Measurements of the forced vital capacity (FVC), the forced expiratory volume in one second (FEV1), the functional residual capacity (FRC), the total lung capacity (TLC) and the residual volume (RV).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Alain Gevenois, MD, PhD, Study Director — Erasme University Hospital
Locations (1):
- Erasme University Hospital, Brussels, Brussels Capital, Belgium

REFERENCES:
- [Background] Rodriguez-Roisin R. Toward a consensus definition for COPD exacerbations. Chest. 2000 May;117(5 Suppl 2):398S-401S. doi: 10.1378/chest.117.5_suppl_2.398s. PMID 10843984
- [Background] Myint PK, Lowe D, Stone RA, Buckingham RJ, Roberts CM. U.K. National COPD Resources and Outcomes Project 2008: patients with chronic obstructive pulmonary disease exacerbations who present with radiological pneumonia have worse outcome compared to those with non-pneumonic chronic obstructive pulmonary disease exacerbations. Respiration. 2011;82(4):320-7. doi: 10.1159/000327203. Epub 2011 May 20. PMID 21597277
- [Background] Hansell DM, Bankier AA, MacMahon H, McLoud TC, Muller NL, Remy J. Fleischner Society: glossary of terms for thoracic imaging. Radiology. 2008 Mar;246(3):697-722. doi: 10.1148/radiol.2462070712. Epub 2008 Jan 14. PMID 18195376
- [Background] Rutschmann OT, Cornuz J, Poletti PA, Bridevaux PO, Hugli OW, Qanadli SD, Perrier A. Should pulmonary embolism be suspected in exacerbation of chronic obstructive pulmonary disease? Thorax. 2007 Feb;62(2):121-5. doi: 10.1136/thx.2006.065557. Epub 2006 Nov 13. PMID 17101737
- [Derived] Hackx M, Ghaye B, Coche E, Muylem AV, Gevenois PA. Severe COPD exacerbation: CT features. COPD. 2015 Feb;12(1):38-45. doi: 10.3109/15412555.2014.903916. Epub 2014 Jun 10. PMID 24914492